CLINICAL TRIAL: NCT02681471
Title: Bipolar Versus Monopolar Resection of Benign Prostate Hyperplasia: A Comparison of the Effects on Plasma Electrolytes, Osmolarity and Hemoglobin
Brief Title: Bipolar Versus Monopolar Resection of Benign Prostate Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Attending Anesthesiologist, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/434-992
Record Dates: First submitted 2016-01-30; First posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Acute Hyponatremia
Keywords: Monopolar; Bipolar; TURP syndrome; hyponatremia
MeSH Terms: conditions — Hyponatremia | interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monopolar TURP (Active Comparator): Patients in Group M (Monopolar) were used monopolar resectoscope (Karl Storz, Tottling, Germany) and 5% Mannitol as an irrigation fluid.
  Interventions: Other: 5% Mannitol; Device: monopolar resectoscope
- Bipolar TURP (Active Comparator): Patients in Group B (Bipolar) were used bipolar resectoscope TURis (OLYMPUS, Tokyo, Japan) and 0,9% Sodium chloride as an irrigation fluid.
  Interventions: Other: 0,9% Sodium chloride; Device: bipolar resectoscope TURis

INTERVENTIONS:
Other: 5% Mannitol — Traditional monopolar TURP was performed by using and irrigation fluid containing 5% mannitol ( Resectisol Eczacibasi-Baxter).
  Other Names: Karl Storz resectoscope
  Arms: Monopolar TURP
Other: 0,9% Sodium chloride — Bipolar TURP was carried out by using a 24 Fr TURis (OLYMPUS) resectoscope and irrigation fluid containing 0,9 % sodium chloride.
  Other Names: TURis (OLYMPUS) resectoscope
  Arms: Bipolar TURP
Device: monopolar resectoscope
  Arms: Monopolar TURP
Device: bipolar resectoscope TURis
  Arms: Bipolar TURP

SUMMARY:
Aim of this prospective clinical study was to compare two different surgical techniques and used solutions on serum electrolytes, bleeding and Transurethral Resection of Prostate (TURP) syndrome undergoing TURP.

Fifty-three patients scheduled for elective TURP were enrolled in this prospective clinical study. Patients were included one of two groups (Group Monopolar and Group Bipolar).

DETAILED DESCRIPTION:
Background and Purpose:

Aim of this prospective clinical study was to compare two different surgical techniques and used solutions on serum electrolytes, bleeding and Transurethral Resection of Prostate (TURP) syndrome undergoing TURP.

Methods:

Fifty-three patients scheduled for elective TURP were enrolled in this prospective clinical study. Patients were divided into two groups. Patients in Group M (Monopolar) (n=25) were used monopolar resectoscope (Karl Storz, Tottling, Germany) and 5% mannitol as irrigating solution. Patients in Group B (Bipolar) (n=25) were used bipolar resectoscope TURis (OLYMPUS, Tokyo, Japan) and isotonic saline as irrigating solution. Patients who received spinal anaesthesia were given 2.5-3 ml 0.5% hyperbaric bupivacain intrathecally and others were given general anaesthesia. Patients demographics, prostate volumes, hemodynamic parameters, volumes of irrigation and IV solutions were recorded. Blood samples were collected preoperatively (control), 45 minutes after the induction (2nd Measurement) and 1 hour after the end of the operation for analyzing serum electrolytes, osmolarity, hemoglobin values.

ELIGIBILITY:
Inclusion Criteria:

* Men were older than 50 years
* Men suffered from symptomatic benign prostatic hyperplasia.

Exclusion Criteria:

* History of severe heart failure
* History of respiratory failure
* History of bleeding diathesis

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Serum sodium level | 0-3 hours
  Sodium level (meq /L)

SECONDARY OUTCOMES:
Serum osmolarity | 0-3 hours
  Osmolarity (mosm/kg)
Serum potassium levels | 0-3 hours
  Potassium level (meq/L)
Serum hemoglobin level | 0-3 hours
  Hemoglobin level (g /dL)

OTHER OUTCOMES:
Systolic blood pressure | 0-3 hours
  mm Hg
Diastolic blood pressure | 0-3 hours
  mm Hg
Heart rate | 0-3 hours
  beat/min

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Savran Karadeniz, MD, Principal Investigator — Istanbul University
Locations (1):
- Meltem Savran Karadeniz, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Michielsen DP, Coomans D, Braeckman JG, Umbrain V. Bipolar transurethral resection in saline: the solution to avoid hyponatraemia and transurethral resection syndrome. Scand J Urol Nephrol. 2010 Sep;44(4):228-35. doi: 10.3109/00365591003720275. PMID 20345336
- [Derived] Karadeniz MS, Bayazit E, Aksoy O, Salviz EA, Tefik T, Sanli O, Sungur MO, Tugrul KM. Bipolar versus monopolar resection of benign prostate hyperplasia: a comparison of plasma electrolytes, hemoglobin and TUR syndrome. Springerplus. 2016 Oct 7;5(1):1739. doi: 10.1186/s40064-016-3407-7. eCollection 2016. PMID 27777873